CLINICAL TRIAL: NCT04099745
Title: Comparing the Accuracy of Different Blood Glucose Monitoring Systems (CGM and FGM) With Venous Blood Glucose
Brief Title: Comparing the Accuracy of Different Blood Glucose Monitoring Systems (CGM and FGM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KY20190823-02
Record Dates: First submitted 2019-09-16; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
Keywords: FGM; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM（continuous glucose monitoring） (Experimental): Each diabetic patient received three CGM tests within 14 days of FGM monitoring, on days 1-3, 6-9 and 12-14, respectively.
  Interventions: Device: CGM
- FGM（Flash glucose monitoring） (Experimental): Each diabetic patient received one FGM test for 14 days.
  Interventions: Device: FGM

INTERVENTIONS:
Device: CGM — Continuous Glucose Monitoring System
  Arms: CGM（continuous glucose monitoring）
Device: FGM — Flash glucose monitoring System
  Arms: FGM（Flash glucose monitoring）

SUMMARY:
To compare the accuracy of different blood glucose monitoring systems (CGM and FGM) in diabetic patients with insufficient islet function.

DETAILED DESCRIPTION:
To compare the accuracy of different blood glucose monitoring systems (CGM and FGM) in diabetic patients with insufficient islet function with Venous Blood Glucose (including FGM early, middle and late, pre-and post-meal, high and low blood glucose).

ELIGIBILITY:
Inclusion Criteria:

* volunteer to participate and be able to sign informed consent prior to the trial.
* patients with type 2 diabetes or type 1 diabetes, aged 18-80 years old.
* No acute complications such as diabetic ketoacidosis, diabetic hyperosmolar syndrome, etc.
* Subjects are able and willing to monitor peripheral blood sugar and regularity of diet and exercise.

Exclusion Criteria:

* Patients with insulin allergy.
* Impaired liver and kidney function with ALT 2.5 times higher than the upper limit of normal value; Serum creatinine was 1.3 times higher than the upper limit of normal.
* Drug abuse and alcohol dependence in the past 5 years.
* Systemic hormone therapy was used in the last three months.
* Patients with poor compliance and irregular diet and exercise.
* Patients with pregnancy, lactation or pregnancy intention.
* Any other obvious conditions or associated diseases determined by the researcher: such as severe cardiopulmonary diseases, endocrine diseases, neurological diseases, tumors and other diseases, other pancreatic diseases, history of mental diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of different blood glucose monitoring systems (CGM and FGM) with intravenous blood glucose level as the gold standard | 2 weeks
  To compare the accuracy of different blood glucose monitoring systems (CGM and FGM) with intravenous blood glucose level as the gold standard in diabetic patients with insufficient islet function.

SECONDARY OUTCOMES:
three-day blood glucose fluctuation of CGM | 3 DAYS
forty-day blood glucose fluctuation of FGM | 14 days

IPD SHARING:
Plan to Share IPD: Undecided